CLINICAL TRIAL: NCT03486171
Title: Quality of Tracheal Intubation in Prehospital Emergency Setting and Measurement of Risk Factors of Difficult Intubation in This Context
Brief Title: Tracheal Intubation and Prehospital Emergency Setting
Acronym: SMURIDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Michel GALINSKI, Principal investigator, University Hospital, Bordeaux
Other Study IDs: CHUBX-URG-01
Record Dates: First submitted 2018-01-24; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Tracheal Intubation Morbidity; Emergency Medicine
Keywords: difficult intubation; prehospital emergency; risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In prehospital emergency setting, tracheal intubation is a frequent procedure (8% of interventions). Its objective is to control and protect upper airways and to optimize ventilation and oxygenation in patients with life-threatening distress. Intubation is a technical procedure which is associated with few difficulties with, in rare cases, the impossibility to do it. There are specificities of the out-of-hospital emergency with some risk factors that have been recognized in this context as well as the impossibility of assessing predictive factors of difficult intubation linked to the patient. The objective of the investigators was to describe the quality of tracheal intubation in prehospital emergency setting.

DETAILED DESCRIPTION:
National and international guidelines have the objective to optimize the airway management modalities and to minimize the risk of complications in relation to this procedure. In contrast to the operating-room where intubation is performed daily in standardized conditions, in prehospital emergency setting, the environment and circumstances are variable and have an impact on the gesture as has been demonstrated. However, there are few studies about this issue, and these one are relatively ancients although that orotracheal intubation procedures in emergency are now well defined and that the algorithms for the management of difficult intubation have been well diffused in the emergency area these last 10 years. The last study about this topic has been published in 2012 involving more than 600 patients included between 2008 and 2010.

Difficult intubation rate, defined with a number of attempts over 2 or the use of an alternative technic was 11%. Another study with more than 2000 patients had found a rate of 6%. A study comparing the intubation difficulty scale score between two types of blades in 800 patients had found a rate of difficult intubation from 9 to 12%. The algorithms of the management of difficult intubation were largely based on the result of studies performed by anesthesiologists in operating ward. The objective will be to describe the quality of intubation and to measure risk factors of difficult intubation. The investigators are going to collect data about all patients intubated in prehospital emergency setting with the objective to measure the difficult intubation rate and to describe variables associated with difficult intubation. The follow up will be restricted to the area of prehospital emergency setting.

ELIGIBILITY:
Inclusion Criteria:

* all patients intubated by Emergency Medical System (EMS) team

Exclusion Criteria:

* none

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with life-threatening distress requiring emergency intubation.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Difficult intubation rate | One hour
  Difficult intubation is defined with an Intubation Difficult Scale score > 5; Intubation Difficult Sale (IDS) is ranged from 0 (easy intubation) to infinity (impossibility to intubate trachea).

SECONDARY OUTCOMES:
Risk factors of difficult intubation | one hour
  Circumstances of intubation (outside/inside), patient on the floor or not, cardiac arrest or not and if yes resuscitation during the intubation or not, nature of the drugs for sedation during rapid sequence induction, pharyngeal or laryngeal hemorrhage.
Patient characteristics | one hour
  sex , age, body mass index, acute disease (trauma or medical), criteria associated with difficult airway access (mouth opening, thyroid-chin distance, neck circumference), pharyngeal or laryngeal tumor.
Events during and after intubation | one hour
  desaturation, vomiting, low blood pressure, tachycardia or bradycardia, cardiac arrest, others.

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL GALINSKI, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU DE BORDEAUX- Hôpital PELLEGRIN - SAMU-SMUR 33, Bordeaux
  - Aphp, Hopital Raymond Poincare - Samu-Smur 92, Garches
  - Ch Garges Les Gonesses, Garges-lès-Gonesse
  - Chu de Grenoble - Samu-Smur 38, Grenoble
  - Ch de Perigueux - Samu-Smur 24, Périgueux